CLINICAL TRIAL: NCT03476499
Title: Near Infrared Imaging for the Assessment of Tissue Viability: Can NIR Images Predict Necrosis?
Brief Title: Near Infrared Imaging and Flap Necrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAPCR ID:18-5013
Record Dates: First submitted 2018-01-29; First posted 2018-03-26 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Flap Necrosis

STUDY DESIGN:
Intervention Model Description: KENT CAMERA MULTISPECTRAL IMAGING DEVICE Health Canada Medical device Licence: 99281 First Issue Date: 2017/06/07 Device class 2 Handheld near infrared multispectral imaging device with custom software. A new commercially available imaging technology uses NIR spectroscopy to measure regional tissue hemoglobin oxygenation, StO2. These images are processed to produce a colour coded StO2 image of a large tissue area (~6" by 4"). Since the image device doesn't contact the skin the depth of measurement is ~2mm instead of ~10mm with a point system. Compared to dye based angiography methods, StO2 NIR imaging does not require the injection of a dye. The advantage of the NIR imaging device over point NIR systems is a lack of patient contact. Thus StO2 NIR imaging is completely non-invasive, non-contact. Images can be captured and displayed in less than 5 seconds therefore imaging can be repeated as needed with no risk to the patient and no cost for disposables.
Masking Description: The physician taking the images will be blinded to the images until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Planned skin flap procedure (Experimental): Inclusion Criteria: i. Planned skin flap procedure, ii. SpO2 above 96% and iii: Written informed consent.
  Exclusion criteria: Use of epinephrine, patent blue V or methelyne blue during procedure.
  The near infrared imaging NIR device is experimental. Experimental means that the NIR imaging is not used routinely in patients' care.
  The research will require no extra study visits. Images will be taken at 3 - 4 time points and a separate photo consent will be obtained prior to imaging.
  * One set of pre-procedure images, NIR images will be taken prior to the start of the breast surgery.
  * One set of intra-operative Images that will be taken intra-operatively following the mastectomy.
  * One to two follow-up sets of NIR images will be taken at the standard post-op follow-up visits at 1 to 2 weeks post-op for up to 30 days post-op. Follow-up visits will be scheduled as per the standard of care.
  Interventions: Device: Near Infrared Imaging (NIR) device

INTERVENTIONS:
Device: Near Infrared Imaging (NIR) device — Handheld near infrared multispectral imaging device with custom software.
  Other Names: KENT CAMERA MULTISPECTRAL IMAGING DEVICE

SUMMARY:
Skin flaps following mastectomy breast surgery that do not have enough oxygen are at risk for necrosis which can increase wound healing problems, postoperative recovery time and be costly to the hospital systems and affect the patient quality of life, poor esthetic results and overall reconstructive success. Mastectomy skin flap necrosis (MSFN) has an incidence of 10-15% with higher rates (7% - 30%) in mastectomy procedures with immediate reconstruction. Intraoperative assessment of the circulation in skin flaps is currently done with clinical assessment tools utilizing somewhat subjective identifiers such as flap color, capillary refill, temperature and dermal edge bleeding to determine the viability of the flap. Several technologies have been developed to assist in the clinical judgement of skin flaps but these technologies are not yet widely used because of the cost of the technology, the time required to image the patient, the intravenous injection of indocyanine green (ICG) dye required for contrast and the inability to image repeatedly and in different environments (pre-op, intra-op and post-op). A new commercially available imaging technology uses NIR spectroscopy to measure regional tissue hemoglobin oxygenation, using images that are taken 12 inches away from the patient. Preclinical data shows that NIR can predict necrosis in flaps but clinical data is needed to characterize and assess the value of the technology in plastic and reconstructive surgery. The purpose of this research study is to explore the ability of NIR imaging to predict skin flap tissue viability in the clinical setting of immediate breast reconstruction procedures. Study Design: This is a prospective, non-interventional study that will explore the ability of NIR imaging to predict of tissue viability in immediate breast reconstruction procedures. Necrosis will be scored using the SKIN score. Participation in the study will not impact patient care; all patients will receive standard care.

DETAILED DESCRIPTION:
Background of the study:

There are commercial medical devices that measure the spectrum of near infrared light reflected from at a single location of tissue. These non-imaging devices are also called point NIR spectroscopy devices. Point NIR spectroscopy devices have been used to monitor blood perfusion to free flaps and mastectomy flaps. The unit of measurement is StO2; StO2 is a measure of hemoglobin oxygen saturation weighted towards the saturation in the microvascular bed as opposed to SaO2 or SvO2 which correspond to the arterial and venous hemoglobin saturation respectively. StO2 is mixed arterial - venous measure of hemoglobin oxygen saturation. Point devices use a light delivery and collection probe that needs to be in contact with tissue. They can measure on the order of ~10mm deep over an area of approximately 1cm by 1cm depending on the configuration of the device. Some studies using point devices have shown significant differences in StO2 values in flaps that became necrotic versus flaps that remained viable. NIR point systems however are not widely used intraoperatively because they need to be brought in contact with the tissue being measured. They also measure small areas thereby necessitating measurements over many spatially distinct points on the flap to get a comprehensive measurement of flap oxygenation.

Rationale for this study A new commercially available imaging technology uses NIR spectroscopy to measure regional tissue hemoglobin oxygenation, StO2. The device is based on the same principles as point NIR spectroscopy devices but instead of contacting the skin a set of images are taken 12 inches away from the patient. These images are processed to produce a colour coded StO2 image of a large tissue area (~6" by 4"). Since the image device doesn't contact the skin the depth of measurement is ~2mm instead of ~10mm with a point system. Compared to dye based angiography methods, StO2 NIR imaging does not require the injection of a dye. The advantage of the NIR imaging device over point NIR systems is a lack of patient contact. Thus StO2 NIR imaging is completely non-invasive, non-contact. Images can be captured and displayed in less than 5 seconds therefore imaging can be repeated as needed with no risk to the patient and no cost for disposables. Preclinical data shows that NIR can predict necrosis in flaps but clinical data is needed to characterize and assess the value of the technology in plastic and reconstructive surgery.

Study hypotheses or research questions This study will explore the ability of NIR imaging to predict of tissue viability in immediate breast reconstruction procedures. Necrosis will be scored using the SKIN score.

Primary objectives and secondary objectives:

Aim 1: To establish the NIR parameters that are consistent with flap viability. Aim 1: To develop parameters to predict flap viability intraoperatively. Aim 3: To determine if NIR values correspond to SKIN scores

Significance of the study The Innovation is a non-contact, non-invasive means to map/image the oxygen available to an area of tissue. It requires no setup time and there are no consumables associated with its measurement method. As cellular respiration in tissue requires an adequate supply of oxygen, the tissue hemoglobin oxygen saturation image provided by the Innovation can detect areas of tissue that are threatened by a poor oxygen supply. The oxygenation measures provided by the device give surgeons insight into the healing potential of skin flaps in procedures such as mastectomies. Skin flaps that are not sufficiently oxygenated are at risk for necrosis which can be costly to the hospital systems and affect the patient quality of life. The Innovation's oxygenation image assists surgeons in identifying areas of flap ischemia intra-operatively and can be used to monitor flaps post-operatively. With early identification of ischemic areas surgeons can intervene earlier to reduce the risk of flap necrosis.

ELIGIBILITY:
Inclusion Criteria:

* i. Planned skin flap procedure
* ii. SpO2 above 96%
* iii: Written informed consent.

Exclusion Criteria:

* Use of epinephrine, patent blue V or methelyne blue during procedure

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Extent of mastectomy skin flap necrosis | 1 month
  Partial/superficial necrosis and full-thickness necrosis as quantified by a SKIN score. These areas will be correlated with the intraoperative StO2 values from the NIR images.

SECONDARY OUTCOMES:
Infection | 1 month
  Superficial, deep or organ space surgical site infection. Patients treated with oral or IV antibiotics will be documented, including patients who have loss of implant due to infection.
Wound Dehiscence or Implant Extrusion | 1 month
  Wound breakdown and/or exposure of implant will be documented.
Seroma/Hematoma | 1 month
  Any evidence of seroma /hematoma will be documented as will any surgical intervention or observation.
Removal or Loss of Implant | 1 month
  Patients who require removal of their implants will be documented along with the reason for removal of implant.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan OP Hofer, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Sinai Health System, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No